CLINICAL TRIAL: NCT03181451
Title: A Phase 1, Open-Label, Randomised, Repeat Dose, Parallel Group Study to Evaluate the PK, Safety, Tolerability of Ferric Maltol at 3 Dosage Levels in Paediatric Subjects Aged 10-17 Years of Age With Iron Deficiency
Brief Title: Evaluate the PK, Safety, Tolerability of Ferric Maltol at 3 Dosage Levels in Paediatric Subjects With Iron Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ST10-01-103
Record Dates: First submitted 2017-05-23; First posted 2017-06-08 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Iron Deficiency, Anaemia in Children; Iron-Deficiency
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — ferric maltol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1:1 ratio and stratified by co-variates for age and sex. This will ensure that a minimum of 25% of each gender and at least 3 children per age group are enrolled in each Ferric Maltol dose group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 mg Ferric Maltol (Active Comparator): 12 subjects will receive 30 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 30mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Interventions: Drug: Ferric Maltol
- 16.6 mg Ferric Maltol (Active Comparator): 12 subjects will receive 16.6 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 16.6mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Interventions: Drug: Ferric Maltol
- 7.8 mg Ferric Maltol (Active Comparator): 12 subjects will receive 7.8 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 7.8mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Interventions: Drug: Ferric Maltol

INTERVENTIONS:
Drug: Ferric Maltol — To assess the pharmacokinetics and iron uptake of Ferric Maltol through measurement of serum iron, transferrin saturation (TSAT) and plasma concentrations of maltol and maltol glucuronide.
  Other Names: ST10; Feraccru

SUMMARY:
The study has been designed to establish the pharmacokinetics (PK) and iron uptake of Ferric Maltol in children and adolescents aged 10-17 years using two (2) lower dose strengths in comparison to the EU-approved 30mg BID dose in adults with IDA in IBD.

DETAILED DESCRIPTION:
Phase I, open label, randomized, repeat dose, multicentre, pharmacokinetic study to assess the Safety and Tolerability of Ferric Maltol in 3 different dosages.

36 eligible patients will be randomized in a 1:1:1 ratio to one of the following 3 dosages for 9 days BID and a single dose on Day 10:

* 30mg ferric maltol capsules
* 16.6 mg ferric maltol capsules
* 7.8 mg ferric maltol capsules

Subject participation in the study will consist of 3 stages:

Screening: up to 14 days Treatment period: 10 days treatment period with 2 visits on Day 1 and Day 10 for PK blood sampling. Patients will be randomly allocated to one of the three Ferric Maltol dose groups according to centralized treatment allocation scheme.

Post-treatment Safety Follow-up:3-10 days following completion of the treatment period or premature discontinuation of study medication

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the information given in the Independent Ethics Committee (IEC) approved Information Sheet and Consent form. The parent or guardian of the study subject must sign and date the informed consent and authorisation to use protected health information (PHI) in accordance with national and local subject privacy regulations prior to any study mandated procedure. The study participant will be asked to provide their assent to participate in the study using the IEC approved Assent form.
2. Willing and able to comply with study requirements.
3. Age ≥10 to ≤17 years at the time of informed consent and throughout duration of the study.
4. A current diagnosis of iron deficiency (with or without anaemia); iron deficiency defined by ferritin <30 µg/L, or ferritin <50 µg/L with transferrin saturation (TSAT) <20%, as measured by the central laboratory at the Screening visit (subjects with or without anaemia may be enrolled providing Hb is ≥8.5 g/dL as measured at the Screening visit).
5. Where appropriate, female subjects of childbearing potential must agree to use a reliable method of contraception until study completion and for at least 4 weeks following their final study visit. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), complete sexual abstinence, a vasectomized partner and oral contraceptive medications.

Exclusion Criteria:

1. Has untreated or untreatable severe malabsorption syndrome e.g., untreated coeliac disease
2. Has received within 28 days prior to Screening intramuscular or intravenous (IV) injection or administration of depot iron preparation.
3. Has received oral iron supplementation within 7 days prior to Screening
4. Has received blood transfusion within 12 weeks prior to Screening or is scheduled to have blood transfusion or donations during the study period.
5. Has concomitant disease that would significantly compromise iron absorption or absorbed iron utilisation such as swallowing disorders and/or extensive small bowel resection.
6. Has chronic renal disease (eGFR <30mL/min), as assessed at Screening based on serum creatinine.
7. Known hypersensitivity or allergy to either the active substance or excipients of Ferric Maltol capsules.
8. Has a known contraindication for treatment with iron preparations, e.g. haemochromatosis, chronic haemolytic disease, sideroblastic anaemia, thalassemia, or lead intoxication induced anaemia.
9. Impaired liver function as indicated by alanine aminotransferase (ALT) or aspartate transaminase (AST)>2.0 times upper normal limit as measured at the Screening visit.
10. Active acute inflammatory disease, including IBD flare or disease exacerbation, which in the opinion of the Investigator, is clinically significant.
11. Active chronic or acute infectious diseases requiring antibiotic treatment.
12. Pregnant or breast feeding.
13. Concomitant medical conditions with extensive active bleeding, other than menstrual cycles; subjects who suffer from menorrhagia may be included at the Investigator's discretion.
14. Scheduled or expected hospitalisation and/or surgery during the course of the study
15. Participation in any other interventional clinical study within 28 days prior to Screening.
16. Cardiovascular, liver, renal, hematologic, psychiatric, neurologic, gastrointestinal, immunologic, endocrine, metabolic, respiratory or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or objectives of the study drug or severely limit the lifespan of the subject.
17. Any other unspecified reason that, in the opinion of the Investigator or the Sponsor make the subject unsuitable for enrolment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 mg Ferric Maltol: 12 subjects will receive 30 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 30 mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Ferric Maltol: To assess the pharmacokinetics and iron uptake of Ferric Maltol through measurement of serum iron, transferrin saturation (TSAT) and plasma concentrations of maltol and maltol glucuronide.
- 16.6 mg Ferric Maltol: 13 subjects will receive 16.6 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 16.6 mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Ferric Maltol: To assess the pharmacokinetics and iron uptake of Ferric Maltol through measurement of serum iron, transferrin saturation (TSAT) and plasma concentrations of maltol and maltol glucuronide.
- 7.8 mg Ferric Maltol: 12 subjects will receive 7.8 mg Ferric Maltol twice daily for 9 days (Days 1-9) plus a final 7.8 mg dose on the morning of Day 10. PK study Day 1 & Day 10.
  Ferric Maltol: To assess the pharmacokinetics and iron uptake of Ferric Maltol through measurement of serum iron, transferrin saturation (TSAT) and plasma concentrations of maltol and maltol glucuronide.
Period: Overall Study
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Started | 12 | 13 | 12
Completed | 12 | 11 | 12
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol | Total
Number analyzed (Participants) | 12 | 13 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.56) | 13.7 (1.80) | 14.2 (2.12) | 14.0 (1.80)
Age, Customized [Count of Participants; unit: Participants]
  10-14 | 8 | 7 | 8 | 23
  15-17 | 4 | 6 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 4 | 5 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 11 | 13 | 11 | 35
  Ethnicity: Unknown | 1 | 0 | 1 | 2
Height [Mean (Standard Deviation); unit: m] | 1.590 (0.0641) | 1.601 (0.855) | 1.618 (0.0914) | 1.603 (0.0799)
Weight [Mean (Standard Deviation); unit: kg] | 57.83 (20.961) | 62.77 (23.330) | 52.07 (9.661) | 57.41 (18.758)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.695 (7.4067) | 24.265 (7.7647) | 19.760 (2.7049) | 22.182 (6.4355)
Haemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.27 (0.856) | 12.75 (1.067) | 12.37 (1.418) | 12.47 (1.124)
Ferritin [Mean (Standard Deviation); unit: μg/L] | 16.2 (7.18) | 18.8 (8.29) | 13.8 (8.34) | 16.3 (8.02)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration [Cmax] of Maltol Glucuronide on Day 1
Description: Descriptive statistics and population PK analysis of maltol glucuronide Cmax from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 2.4518 (1.29590) | 1.1632 (0.18435) | 0.5299 (0.02245)

2. Primary Outcome: Maximum Plasma Concentration [Cmax] of Maltol Glucuronide on Day 10
Description: Descriptive statistics and population PK analysis of maltol glucuronide Cmax from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 4.2355 (0.78110) | 2.1028 (0.13342) | 0.9926 (0.02349)

3. Primary Outcome: Area Under The Curve [AUC] of Maltol Glucuronide on Day 1
Description: Descriptive statistics and population PK analysis of maltol glucuronide AUC from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h*mg/L | 11.090 (3.9033) | 5.613 (0.7589) | 2.585 (0.0968)

4. Primary Outcome: Area Under The Curve [AUC] of Maltol Glucuronide on Day 10
Description: Descriptive statistics and population PK analysis of maltol AUC from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h*mg/L | 20.511 (1.7997) | 10.518 (0.5277) | 5.016 (0.1133)

5. Primary Outcome: Average Plasma Concentration [Cave(0-6h)] of Maltol Glucuronide on Day 10
Description: Descriptive statistics and population PK analysis of maltol glucuronide Cave(0-6h) from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 3.4186 (0.29995) | 1.7531 (0.08795) | 0.8360 (0.01889)

6. Primary Outcome: Time of Maximum Plasma Concentration [Tmax] of Maltol Glucuronide on Day 1
Description: Descriptive statistics and population PK analysis of maltol glucuronide Tmax from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h | 1.00 [0.75 to 1.00] | 1.00 [0.75 to 1.00] | 1.00 [1.00 to 1.00]

7. Primary Outcome: Time of Maximum Plasma Concentration [Tmax] of Maltol Glucuronide on Day 10
Description: Descriptive statistics and population PK analysis of maltol glucuronide Tmax from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h | 0.75 [0.75 to 0.75] | 0.75 [0.75 to 0.75] | 0.75 [0.75 to 0.75]

8. Primary Outcome: Half Life [t1/2] of Maltol Glucuronide on Day 1
Description: Descriptive statistics and population PK analysis of maltol glucuronide t1/2 from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h | 11.384 (5.4738) | 10.447 (1.8503) | 10.806 (0.4707)

9. Primary Outcome: Ratio of Maximum Plasma Concentration [Cmax] of Maltol Glucuronide on Day 10/Day 1
Description: Descriptive statistics of ratio maltol glucuronide Cmax Day 10/Day 10 from PK samples collected on Day 1 and Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 and Day 10, pre-dose and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
ratio | 1.956 (0.6210) | 1.836 (0.2109) | 1.875 (0.0537)

10. Primary Outcome: Ratio of Area Under The Curve [AUC] of Maltol Glucuronide on Day 10/Day 1
Description: Descriptive statistics of ratio maltol glucuronide AUC Day 10/Day 10 from PK samples collected on Day 1 and Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 and Day 10, pre-dose and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
ratio | 2.030 (0.6695) | 1.899 (0.2286) | 1.942 (0.0582)

11. Primary Outcome: Average Serum Concentration [Cave(0-6h)] of Iron on Day 10
Description: Descriptive statistics and population PK analysis of iron Cave(0-6h) from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 1.1667 (0.61420) | 0.9557 (0.29645) | 0.9748 (0.39783)

12. Primary Outcome: Change From Pre-Dose (Ctrough) to Maximum Post-Dose (Cmax) in Serum Iron on Day 1
Description: Descriptive statistics and population PK analysis of change in serum iron [Ctrough to Cmax] from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 0.6159 (0.32320) | 0.4102 (0.22144) | 0.21715 (0.11873)

13. Primary Outcome: Change From Pre-Dose (Ctrough) to Maximum Post-Dose (Cmax) in Serum Iron on Day 10
Description: Descriptive statistics and population PK analysis of change in serum iron [Ctrough to Cmax] from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 11
mg/L | 0.5486 (0.32367) | 0.3625 (0.15333) | 0.2251 (0.08362)

14. Primary Outcome: Pre-dose Adjusted Incremental Area Under the Curve [AUC(0-6h)] of Serum Iron on Day 1
Description: Descriptive statistics and population PK analysis of pre-dose adjusted incremental AUC(0-6h) of serum iron from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h*mg/L | 6.711 (2.5721) | 5.963 (1.7793) | 3.928 (1.1318)

15. Primary Outcome: Pre-dose Adjusted Incremental Area Under the Curve [AUC(0-6h)] of Serum Iron on Day 10
Description: Descriptive statistics and population PK analysis of pre-dose adjusted incremental AUC(0-6h) of serum iron from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 11
h*mg/L | 7.000 (3.6852) | 5.734 (1.7787) | 5.849 (2.3870)

16. Primary Outcome: Pre-dose Adjusted Incremental Area Under the Curve [AUC(0-6h)] of Transferrin Saturation (TSAT) on Day 1
Description: Descriptive statistics and population PK analysis of pre-dose adjusted incremental AUC(0-6h) of TSAT from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h*% | 179.47 (60.259) | 159.21 (50.723) | 104.50 (41.009)

17. Primary Outcome: Pre-dose Adjusted Incremental Area Under the Curve [AUC(0-6h)] of Transferrin Saturation (TSAT) on Day 10
Description: Descriptive statistics and population PK analysis of pre-dose adjusted incremental AUC(0-6h) of TSAT from PK samples collected on Day 10. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: h*%
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 11
h*% | 180.14 (76.193) | 149.40 (37.799) | 157.43 (81.693)

18. Primary Outcome: Apparent Systemic Clearance (CL/F) of Iron on Day 1
Description: Descriptive statistics and population PK analysis of serum iron CL/F from PK samples collected on Day 1
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
L/h | 1.321 (0.6945) | 0.654 (0.2441) | 0.324 (0.1517)

19. Primary Outcome: Apparent Systemic Clearance (CL/F) of Iron on Day 10
Description: Descriptive statistics and population PK analysis of serum iron CL/F from PK samples collected on Day 10
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 11
L/h | 3.264 (2.2297) | 1.757 (0.6673) | 0.808 (0.3089)

20. Primary Outcome: Apparent Volume of Distribution (V/F) of Iron on Day 1
Description: Descriptive statistics and population PK analysis of iron V/F from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
L | 22.114 (7.2315) | 14.244 (4.8083) | 10.462 (3.1033)

21. Primary Outcome: Apparent Volume of Distribution (V/F) of Transferrin Saturation (TSAT) on Day 1
Description: Descriptive statistics and population PK analysis of TSAT V/F from PK samples collected on Day 1
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: As PPD analysis was performed, the V/F could not be estimated.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

22. Primary Outcome: Apparent Volume of Distribution (V/F) of Transferrin Saturation (TSAT) on Day 10
Description: Descriptive statistics and population PK analysis of TSAT V/F from PK samples collected on Day 10
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: As PPD analysis was performed, the V/F could not be estimated.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

23. Primary Outcome: Ratio Auc(0-6) Maltol Glucuronide Day 10/Day 1
Description: Ratio AUC0-6h measured after last dose of Ferric Maltol on Day 10 vs first dose Day 1.
Time Frame: Day 1 to Day 10 (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
Ratio | 1.942 (0.0582) | 1.899 (0.2286) | 2.030 (0.6695)

24. Primary Outcome: Serum Iron - RAUC(0-6h) D10/D1
Description: Serum Iron - RAUC(0-6h) Day 10/Day 1
Time Frame: Measured after first and last dose of Ferric Maltol on Day 1 & Day 10 (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 12
Ratio | 1.529 (1.4673) | 1.020 (0.3170) | 1.038 (0.3973)

25. Primary Outcome: Transferrin Saturation (%) Day 1, Baseline
Description: Transferrin Saturation (TSAT%) Day 1, baseline
Time Frame: Measured after first dose of Ferric Maltol on Day 1 (0h)
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage saturation
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
percentage saturation | 11.5 (5.66) | 16.8 (9.25) | 15.8 (9.31)

26. Primary Outcome: Transferrin Saturation (%) Day 1, Maximum Response (%)
Description: Transferrin Saturation (TSAT%) Day 1, maximum response (%)
Time Frame: Measured after first dose of Ferric Maltol on Day 1 (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage saturation
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
percentage saturation | 18.68 (7.13) | 28.261 (8.4784) | 32.845 (10.5913)

27. Primary Outcome: Transferrin Saturation Day 1, Time to Maximum Response Tmax
Description: Transferrin Saturation (TSAT%) Day 1, time to maximum response Tmax (h). Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Measured after first dose of Ferric Maltol on Day 1. (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Median (Full Range); unit: hour
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
hour | 4.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [3.00 to 5.00]

28. Primary Outcome: Transferrin Saturation (%) Day 10, Maximum Response (%)
Description: Transferrin Saturation (TSAT%) Day 10, maximum response (%). Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Measured after last dose of Ferric Maltol on Day 10. (0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage saturation
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 12
percentage saturation | 27.779 (13.863) | 27.214 (6.699) | 33.524 (13.633)

29. Primary Outcome: Transferrin Saturation Day 10, Time to Maximum Response Tmax
Description: as for outcome 27
Time Frame: Measured after first dose of Ferric Maltol on Day 10. (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h).
Population: ITT
Measure: Median (Full Range); unit: hour
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 12
hour | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00] | 3.00 [0.00 to 4.00]

30. Primary Outcome: AUC0-inf Day 1 for Maltol Glucuronide
Description: AUC0-inf for Maltol Glucuronide from PK samples collected on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Measured after first dose of Ferric Maltol on Day 1 (0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: h.mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h.mg/L | 8.590 (0.2025) | 17.862 (0.9328) | 34.372 (4.5052)

31. Primary Outcome: AUC0-tau Day 10 for Maltol Glucuronide
Description: AUC0-tau for Maltol Glucuronide from PK samples collected on Day 10. Area under the plasma concentration versus time curve from time 0 to tau.
Time Frame: Measured after last dose of Ferric Maltol on Day 10. (0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: h mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
h mg/L | 8.59 (0.2024) | 17.862 (0.9327) | 34.368 (4.4981)

32. Primary Outcome: Cthrough for Maltol Glucuronide Day 10
Description: Change from pre-dose to last PK samples collected on Day 10 for maltol glucuronide.Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 10 pre-dose to last (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 0.4804 (0.01639) | 0.9762 (0.10586) | 1.8496 (0.67761)

33. Primary Outcome: Serum Iron Cmax Day 1
Description: Maximum serum concentration of serum iron on Day 1. Each subject had 1 pre-dose (0h) and 2 post dose PK blood sampling between (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h). Subjects were assigned to PK blood sampling schedule. For each individual subject the PK blood sampling schedule was the same on Day 1 and Day 10.
Time Frame: Day 1 (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 0.7030 (0.19765) | 1.681 (0.30405) | 1.2328 (0.47471)

34. Primary Outcome: Serum Iron Cmax on Day 10
Description: Maximum serum concentration of serum iron on Day 10.
Time Frame: Day 10 (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 12
mg/L | 1.0338 (0.4023) | 1.0462 (0.3221) | 1.3034 (0.6741)

35. Primary Outcome: Plasma Maltol Glucuronide Cthrough D10/Day1
Description: Minimum concentration between dose time and dose time+TAU
Time Frame: Day 10 (0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
mg/L | 0.4804 (0.0163) | 0.9762 (0.105) | 1.8496 (0.677)

36. Primary Outcome: Apparent Systemic Clearance (CL/F) of Transferrin Saturation (TSAT) on Day 1
Description: Descriptive statistics and population PK analysis of serum TSAT CL/F from PK samples collected on Day 1
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h
Population: As PPD analysis was performed the CL/F could not be estimated.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

37. Primary Outcome: Apparent Systemic Clearance (CL/F) of Transferrin Saturation (TSAT) on Day 10
Description: Descriptive statistics and population PK analysis of serum TSAT CL/F from PK samples collected on Day 10
Time Frame: Day 10 pre-final dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h)
Population: As PPD analysis was performed, the V/F could not be estimated.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Transferrin - Change From Baseline to Day 10, Predose
Description: Change calculated as difference in values measured at Day 1, predose (Baseline) and on Day 10, predose
Time Frame: Day 1 pre-dose to Day 10 pre-dose (0h on each day)
Population: ITT. Only subjects who had baseline samples taken on each PK day.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 11
g/L | -0.085 (0.1510) | -0.147 (0.1419) | 0.032 (0.2275)

39. Secondary Outcome: Ferritin - Change From Baseline to Day 10, Predose
Description: Change calculated as difference in values measured at Day 1, predose (Baseline) and on Day 10, predose.
Time Frame: Pre-dose on Day 1 to Day 10 (0h)
Population: ITT. Only subjects who had baseline samples taken on each PK day.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 11
μg/L | 7.3 (8.22) | 4.1 (3.73) | 0.5 (4.95)

40. Secondary Outcome: Total Iron Binding Capacity - Change From Day 1 to Day 10, Predose
Description: Change calculated as difference in values measured at Day 1, predose and on Day 10, predose
Time Frame: Predose from Day 1 to Day 10 (0h on each day)
Population: ITT. Only subjects who had baseline samples taken on each PK day.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 11
umol/L | -2.12 (3.406) | -3.11 (3.201) | 1.13 (4.452)

41. Secondary Outcome: UIBC - Change From Day 1 to Day 10, Predose
Description: Change calculated as difference in values measured at Day 1, predose and on Day 10, predose
Time Frame: Pre-dose on Day 1 to Day 10 (0h each day)
Population: ITT
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 11 | 11 | 11
umol/L | -2.10 (7.775) | -2.33 (5.525) | -4.49 (8.343)

42. Secondary Outcome: Negative and Positive NTBI Tests on Day 1
Description: Negative and Positive Non-Transferrin Bound Iron [NTBI] tests on Day 1, predose
Time Frame: Day 1 (0h)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
Participants
  Positive | 0 | 0 | 0
  Negative | 12 | 13 | 12

43. Secondary Outcome: Change From Baseline to Day 10 in Haemoglobin Concentration
Description: Change calculated as difference in values measured at Screening (Baseline) and on Day 10
Time Frame: Screening and Day 10 (1-4 hours post-dose)
Population: Safety population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 11
g/dL | -0.03 (0.789) | -0.33 (1.097) | -0.45 (0.301)

44. Secondary Outcome: Change From Baseline to Day 10 in Absolute Reticulocyte Count
Description: Change from Baseline to Day 10 in Absolute Reticulocyte Count collected from PK samples
Time Frame: Change calculated as difference in values measured at Screening (Baseline) and on Day 10.
Population: ITT. Only subjects who had baseline samples and Day 10 samples taken.
Measure: Mean (Standard Deviation); unit: cells*10^12/L
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 5 | 10 | 5
cells*10^12/L | 0.036 (0.0114) | -0.001 (0.0218) | 0.016 (0.0358)

45. Secondary Outcome: Treatment-emergent Adverse Events (AEs) Leading to Premature Discontinuation of Study Drug/PK Assessments
Description: Descriptive summary of incidence and causal relationship of treatment-emergent adverse events leading to discontinuation of study drug/PK assessments according to MedDRA preferred term (PT) and system organ class (SOC)
Time Frame: From first dose of Ferric Maltol on Day 1 through study completion, on average 4 weeks
Population: screened population
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
Participants | 0 | 1 | 0

46. Secondary Outcome: Changes in 12-lead ECG Parameters From Screening to Day 10
Description: Overall clinical interpretation of routine ECG parameters from Screening to Day 10
Time Frame: Screening and Day 10 (1-4 hours post-dose)
Population: Safety population. Subjects who had ECG performed at both visits.
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 10 | 11 | 12
Participants
  Normal | 10 | 11 | 12
  Abnormal | 0 | 0 | 0

47. Secondary Outcome: Concomitant Medications
Description: Number of subjects with concomitant medications Taken by >5% of Subjects
Time Frame: Screening, Day 1, Day 10 and Post-Study Follow-up visit, on average 4 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
Participants | 8 | 13 | 10

48. Secondary Outcome: Negative and Positive NTBI Tests on Day 10, Predose
Description: Negative and Positive Non-Transferrin Bound Iron [NTBI] tests on Day 10, predose
Time Frame: Day 10
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 12 | 11 | 10
Participants
  Positive | 1 | 0 | 0
  Negative | 11 | 11 | 10

49. Secondary Outcome: Treatment-emergent Serious Adverse Event (TESAE)
Description: Descriptive summary of TESAE according to MedDRA preferred Term
Time Frame: From first dose of ferric maltol Day 1 through study completions, on average 4 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 7.8 mg Ferric Maltol | 16.6 mg Ferric Maltol | 30 mg Ferric Maltol
Number analyzed (Participants) | 12 | 13 | 12
Participants | 0 | 0 | 0

50. Primary Outcome: Apparent Systemic Clearance (CL/F) of Maltol Glucuronide on Day 1
Description: Descriptive statistics and population PK analysis of plasma maltol glucuronide CL/F from PK samples collected on Day 1.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h
Population: The dose of maltol glucuronide was not calculable using non-compartmental analysis.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

51. Primary Outcome: Apparent Systemic Clearance (CL/F) of Maltol Glucuronide on Day 10
Description: Descriptive statistics and population PK analysis of plasma maltol glucuronide CL/F from PK samples collected on Day 10.
Time Frame: Day 1 pre-first dose of Ferric Maltol and up to 6 hours post-dose (0h, 0.5-1h, 1-2h, 2-3h, 3-4h, 4-6h
Population: The dose of maltol glucuronide was not calculable using non-compartmental analysis.
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | 30 mg Ferric Maltol | 16.6 mg Ferric Maltol | 7.8 mg Ferric Maltol
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 7/13 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 30 mg Ferric Maltol (N=12) | 16.6 mg Ferric Maltol (N=13) | 7.8 mg Ferric Maltol (N=12)
Palpitations (Cardiac disorders) | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nevus haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03181451/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03181451/SAP_001.pdf